CLINICAL TRIAL: NCT05026710
Title: Better Lithotripsy and Ureteroscopy Evaluation of Stenting (BLUES) A Pragmatic Randomized Multi-center Comparative Effectiveness Study
Brief Title: Better Lithotripsy and Ureteroscopy Evaluation of Stenting (BLUES)
Acronym: BLUES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Coloplast A/S (Industry)
Responsible Party: Principal Investigator, Khurshid Ghani, Associate Professor of Urology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00199486
Record Dates: First submitted 2021-08-23; First posted 2021-08-30 (Actual); Results first posted 2025-10-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Renal Stone; Ureteral Stone
Keywords: Ureteral stent; Ureteroscopy; Lithotripsy
MeSH Terms: conditions — Nephrolithiasis; Ureterolithiasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Silicone (Coloplast Imajin Hydro) ureteral stent (Experimental)
  Interventions: Device: Silicone (Coloplast Imajin Hydro) ureteral stent
- Non-silicone (Polyurethane/Percuflex) ureteral stent (any manufacturer). (Experimental)
  Interventions: Device: Non-silicone (Polyurethane/Percuflex) ureteral stent (any manufacturer)

INTERVENTIONS:
Device: Silicone (Coloplast Imajin Hydro) ureteral stent — During the end of the standard of care ureteroscopy the silicone stent will be placed.
  Arms: Silicone (Coloplast Imajin Hydro) ureteral stent
Device: Non-silicone (Polyurethane/Percuflex) ureteral stent (any manufacturer) — During the end of the standard of care ureteroscopy the Non-silicone (Polyurethane/Percuflex) stent will be placed.
  Arms: Non-silicone (Polyurethane/Percuflex) ureteral stent (any manufacturer).

SUMMARY:
This multi-center trial is being completed to compare patient outcomes related to the Imajin silicone stent in comparison to non-silicone polyurethane stents after ureteroscopy.

Eligible participants will be enrolled and randomly assigned to receive the Imajin silicone stent or a non-silicone stent. In addition, the participants will complete questionnaires and have follow-up information collected (approximately 60 days after surgery).

The trial hypothesizes that a ureteral stent made of silicone, will have superior outcomes when compared to non-silicone stents.

ELIGIBILITY:
Inclusion Criteria:

* Stated willingness to comply with all study procedures and availability for the duration of the study
* Diagnosed with unilateral renal and/or ureteral stones with the largest less than or equal to (≤)2.0 cm in size measured on abdominal x-ray, Ultrasound or computerized tomography (CT) scan

  * Renal stone defined as only renal location of stone(s).
  * Ureteral stone defined as ureteral only or ureteral and renal stone(s).
* Planned unilateral ureteroscopy with stent placement without stent string.
* Ability to take oral medication.
* Ability and willingness to complete and adhere to survey questions and responses throughout study duration.

Exclusion Criteria:

* Known planned secondary or staged procedure
* Presence of anatomical anomalies (for example (e.g.) solitary, horseshoe, fused crossed ectopia, pelvic kidney)
* Presence of any prior urinary diversion (e.g. ileal conduit, orthotopic neobladder)
* Presence of any indwelling ureteral stent prior to ureteroscopy
* Presence of any indwelling nephrostomy tube prior to ureteroscopy
* Ancillary ureteroscopy to treat residual fragments after percutaneous renal stone surgery
* Renal stone located in calyceal diverticulum
* No indication for stent placement (e.g. spontaneous passage)
* Bladder stone location.
* Pregnancy or lactation
* Known allergic reactions to polyurethane or silicone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Khurshid Ghani, MD, MS, FRCS, Principal Investigator — University of Michigan
Locations (10):
- United States (10):
  - Michigan Medicine, Ann Arbor, Michigan
  - Michigan Medicine, Brighton, Michigan
  - Chelsea Hospital (Saint Joseph Mercy), Chelsea, Michigan
  - Henry Ford Macomb Hospital, Clinton Township, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Hospital (Comprehensive Urology), Novi, Michigan
  - William Beaumont Hospital (Michigan Institute of Urology), Royal Oak, Michigan
  - William Beaumont Hospital (Michigan Institute of Urology), Troy, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Integrated Healthcare Association (IHA) (Saint Joseph Mercy Hospital), Ypsilanti, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Becker REN, DiBianco JM, Higgins AM, Konheim J, Kleer E, Leavitt D, King A, Kachroo N, Majdalany SE, Gandham D, Fernandez Moncaleano G, Conrado B, Shoemaker E, Daignault-Newton S, Dauw CA, Ghani KR. Daily Ecological Momentary Assessments of Pain and Ability to Work After Ureteroscopy and Stenting. J Endourol. 2024 Jun;38(6):545-551. doi: 10.1089/end.2023.0625. PMID 38545762

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For the purposes of this trial, enrollment was defined as those who were randomized, remained eligible prior to stent placement, and received the study intervention.
Period: Overall Study
Arm/Group | Silicone (Coloplast Imajin Hydro) Ureteral Stent | Non-silicone (Polyurethane/Percuflex) Ureteral Stent (Any Manufacturer).
Started | 110 | 109
Completed | 107 | 108
Not Completed | 3 | 1
Not completed — No longer met eligibility criteria | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Silicone (Coloplast Imajin Hydro) Ureteral Stent | Non-silicone (Polyurethane/Percuflex) Ureteral Stent (Any Manufacturer). | Total
Number analyzed (Participants) | 110 | 109 | 219
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [50 to 67] | 59 [50 to 67] | 59 [50 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 57 | 116
  Male | 51 | 52 | 103
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasion | 95 | 94 | 189
  African American | 4 | 8 | 12
  Other | 2 | 1 | 3
  Unknown/Refused | 5 | 5 | 10
  Asian | 4 | 1 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic | 101 | 100 | 201
  Hispanic | 0 | 2 | 2
  Unknown/refused | 9 | 7 | 16
Stone Location [Count of Participants; unit: Participants] — Kidney stone location for renal only versus ureteral
  Participants
    Renal Only | 59 | 59 | 118
    Ureter/Ureter + Renal | 48 | 49 | 97
    Withdrawn due to ineligibility | 3 | 1 | 4
Stone Size [Median (Inter-Quartile Range); unit: mm] — Size of stone in millimeters
  mm | 8 [6.3 to 11] | 9 [7 to 11] | 9 [7 to 11]
PROMIS Pain Intensity [Median (Inter-Quartile Range); unit: units on a scale] — This is a 3-item survey which participants select a response for each item from 1=no pain to 5=very severe for intensity of their pain. The sum of responses is then converted into a T-score that ranges from 36.3 to 81.8, with higher scores indicating worse pain intensity. Change is defined as the difference in T-score from baseline to 7-10 days after surgery. Population: *missing baseline PROMIS Pain Intensity due to non-response.
  units on a scale
    number analyzed (Participants) | 106 | 107 | 213
    (all) | 51.4 [36.3 to 61.9] | 54.8 [47.5 to 64.9] | 54.8 [43.1 to 64.9]
PROMIS Pain Interference [Median (Inter-Quartile Range); unit: units on a scale] — This is a 6-item survey which participants select a response for each item from 1=not at all to 5=very much for how much pain interfered with their life. The sum of responses is then converted into a T-score that ranges from 41.0 to 78.3, with higher scores indicating worse pain interference. Change is defined as the difference in T-score from baseline to 7-10 days after surgery. Population: *missing baseline PROMIS Pain Interference due to non-response
  units on a scale
    number analyzed (Participants) | 105 | 107 | 212
    (all) | 56.1 [41.0 to 65.5] | 59.1 [48.5 to 66.4] | 57.1 [41.0 to 66.0]
LURN SI-10 Baseline Measures [Median (Inter-Quartile Range); unit: units on a scale] — The LURN SI-10 (10-Item LURN Symptom Index) assesses urinary frequency, nocturia, urgency, incontinence, bladder pain, voiding and post-micturition symptoms. Responses for each item range from 0 to 4 or 0 to 3 and are then summed for total scores ranging from 0 to 38 (higher scores = worse symptoms/bother). Change is defined as the difference in LURN SI-10 total score from baseline to 7-10 days after surgery. Population: *missing baseline LURN SI-10 due to non-response.
  units on a scale
    number analyzed (Participants) | 106 | 107 | 213
    (all) | 8 [4 to 11] | 7 [5 to 12] | 7 [4 to 11]

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient-Reported Outcomes Measurement Information System (PROMIS®) Scores of Pain-intensity at 7 to 10 Days
Description: This is a 3-item survey which participants select a response for each item from 1=no pain to 5=very severe for intensity of their pain. The sum of responses is then converted into a T-score that ranges from 36.3 to 81.8, with higher scores indicating worse pain intensity. Change is defined as the difference in T-score from baseline to 7-10 days after surgery.
Time Frame: Baseline, 7 to 10 days: Participants can fill out the survey at any time between 7 to 10 days after surgery.
Population: Participants were only included in the analysis if they completed both the baseline survey and the follow-up survey
Measure: Mean (97.5% Confidence Interval); unit: T-score
Arm/Group | Silicone (Coloplast Imajin Hydro) Ureteral Stent | Non-silicone (Polyurethane/Percuflex) Ureteral Stent (Any Manufacturer).
Number analyzed (Participants) | 98 | 96
T-score | 4.28 [1.26 to 7.29] | 2.92 [-0.07 to 5.91]
Statistical Analysis 1: Comparison: Silicone (Coloplast Imajin Hydro) Ureteral Stent vs Non-silicone (Polyurethane/Percuflex) Ureteral Stent (Any Manufacturer); Test type: Superiority; p = 0.26, Regression, Linear

2. Primary Outcome: Change in Patient-Reported Outcomes Measurement Information System (PROMIS®) Scores of Pain-interference at 7 to 10 Days
Description: This is a 6-item survey which participants select a response for each item from 1=not at all to 5=very much for how much pain interfered with their life. The sum of responses is then converted into a T-score that ranges from 41.0 to 78.3, with higher scores indicating worse pain interference. Change is defined as the difference in T-score from baseline to 7-10 days after surgery.
Time Frame: Baseline, 7 to 10 days: Participants can fill out the survey at any time between 7 to 10 days after surgery.
Population: Participants were only included in the analysis if they completed both the baseline survey and the follow-up survey.
Measure: Mean (97.5% Confidence Interval); unit: T-Score
Arm/Group | Silicone (Coloplast Imajin Hydro) Ureteral Stent | Non-silicone (Polyurethane/Percuflex) Ureteral Stent (Any Manufacturer).
Number analyzed (Participants) | 98 | 96
T-Score | 4.62 [1.76 to 7.47] | 3.24 [0.23 to 6.24]
Statistical Analysis 1: Comparison: Silicone (Coloplast Imajin Hydro) Ureteral Stent vs Non-silicone (Polyurethane/Percuflex) Ureteral Stent (Any Manufacturer); Test type: Superiority; p = 0.57, Regression, Linear

3. Secondary Outcome: Change in Patient-Reported Outcomes Measurement Information System (PROMIS®) Scores of Pain-intensity at 4 to 6 Weeks
Description: This is a 3-item survey which participants select a response for each item from 1=no pain to 5=very severe for intensity of their pain. The sum of responses is then converted into a T-score that ranges from 36.3 to 81.8, with higher scores indicating worse pain intensity. Change is defined as the difference in T-score from baseline to 4-6 weeks after surgery.
Time Frame: Baseline, 4 to 6 weeks: Participants can fill out the survey at any time between 4 to 6 weeks after surgery.
Population: Participants were only analyzed for this outcome if the completed the baseline, 7-10 day, and 4-6 week questionnaires
Measure: Mean (95% Confidence Interval); unit: T-Score
Arm/Group | Silicone (Coloplast Imajin Hydro) Ureteral Stent | Non-silicone (Polyurethane/Percuflex) Ureteral Stent (Any Manufacturer).
Number analyzed (Participants) | 93 | 85
T-Score | -6.60 [-9.40 to -3.79] | -9.93 [-13.10 to -6.76]
Statistical Analysis 1: Comparison: Silicone (Coloplast Imajin Hydro) Ureteral Stent vs Non-silicone (Polyurethane/Percuflex) Ureteral Stent (Any Manufacturer); Test type: Superiority; p = 0.58, Regression, Linear

4. Secondary Outcome: Change in Patient-Reported Outcomes Measurement Information System (PROMIS®) Scores of Pain-interference at 4 to 6 Weeks
Description: This is a 6-item survey which participants select a response for each item from 1=not at all to 5=very much for how much pain interfered with their life. The sum of responses is then converted into a T-score that ranges from 41.0 to 78.3, with higher scores indicating worse pain interference. Change is defined as the difference in T-score from baseline to 4-6 weeks after surgery.
Time Frame: Baseline, 4 to 6 weeks: Participants can fill out the survey at any time between 4 to 6 weeks after surgery.
Population: Participants were only analyzed for this outcome if the completed the baseline, 7-10 day, and 4-6 week questionnaires
Measure: Mean (95% Confidence Interval); unit: T-Score
Arm/Group | Silicone (Coloplast Imajin Hydro) Ureteral Stent | Non-silicone (Polyurethane/Percuflex) Ureteral Stent (Any Manufacturer).
Number analyzed (Participants) | 93 | 85
T-Score | -6.38 [-9.18 to -3.58] | -8.08 [-11.29 to -4.87]
Statistical Analysis 1: Comparison: Silicone (Coloplast Imajin Hydro) Ureteral Stent vs Non-silicone (Polyurethane/Percuflex) Ureteral Stent (Any Manufacturer); Test type: Superiority; p = 0.72, Regression, Linear

5. Secondary Outcome: Change in National Institutes of Health (NIH) Lower Urinary Tract Dysfunction Research Network (LURN) Symptoms Index (SI)-10 Scores at 7 to 10 Days
Description: The LURN SI-10 (10-Item LURN Symptom Index) assesses urinary frequency, nocturia, urgency, incontinence, bladder pain, voiding and post-micturition symptoms. Responses for each item range from 0 to 4 or 0 to 3 and are then summed for total scores ranging from 0 to 38 (higher scores = worse symptoms/bother). Change is defined as the difference in LURN SI-10 total score from baseline to 7-10 days after surgery.
Time Frame: Baseline, 7 to 10 days: Participants can fill out the survey at any time between 7 to 10 days after surgery.
Population: Participants were only included in the analysis if they completed both the baseline survey and the day 7-10 follow-up survey
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Silicone (Coloplast Imajin Hydro) Ureteral Stent | Non-silicone (Polyurethane/Percuflex) Ureteral Stent (Any Manufacturer).
Number analyzed (Participants) | 98 | 96
units on a scale | 2.53 [1.42 to 3.64] | 2.90 [1.69 to 4.12]
Statistical Analysis 1: Comparison: Silicone (Coloplast Imajin Hydro) Ureteral Stent vs Non-silicone (Polyurethane/Percuflex) Ureteral Stent (Any Manufacturer); Test type: Superiority; p = 0.50, Mixed Models Analysis

6. Secondary Outcome: Change in NIH LURN SI-10 Scores at 4 to 6 Weeks
Description: The LURN SI-10 (10-Item LURN Symptom Index) assesses urinary frequency, nocturia, urgency, incontinence, bladder pain, voiding and post-micturition symptoms. Responses for each item range from 0 to 4 or 0 to 3 and are then summed for total scores ranging from 0 to 38 (higher scores = worse symptoms/bother). Change is defined as the difference in LURN SI-10 total score from baseline to 4-6 weeks after surgery.
Time Frame: : Baseline, 4 to 6 weeks: Participants can fill out the survey at any time between 4 to 6 weeks after surgery. Baseline, 4 to 6 weeks: Participants can fill out the survey at any time between 4 to 6 weeks after surgery.
Population: Participants were only analyzed for this outcome if the completed the baseline, 7-10 day, and 4-6 week questionnaires
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Silicone (Coloplast Imajin Hydro) Ureteral Stent | Non-silicone (Polyurethane/Percuflex) Ureteral Stent (Any Manufacturer).
Number analyzed (Participants) | 93 | 85
units on a scale | -2.54 [-3.56 to -1.52] | -3.23 [-4.36 to -2.10]
Statistical Analysis 1: Comparison: Silicone (Coloplast Imajin Hydro) Ureteral Stent vs Non-silicone (Polyurethane/Percuflex) Ureteral Stent (Any Manufacturer); Test type: Superiority; p = 0.80, Mixed Models Analysis; Linear mixed effects; covariates: days since URS, study arm, days*arm, baseline LURN, stone location; random intercept with unstructured covariance

7. Secondary Outcome: Composite Healthcare Utilization Metric Within 30 Days (WinRatio)
Description: WinRatio composite healthcare utilization score ranges from 0 to 5 based on each participants highest level of healthcare utilization, with higher score indicating a worse outcome: 0=no HCU, 1=phone call or EMR message, 2=office visit, 3= Emergency Department visit, 4=Unplanned Hospitalization, 5=Hospitalization with ICU care
Time Frame: up to 30 days
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Silicone (Coloplast Imajin Hydro) Ureteral Stent | Non-silicone (Polyurethane/Percuflex) Ureteral Stent (Any Manufacturer).
Number analyzed (Participants) | 107 | 108
units on a scale | 0 [0 to 1] | 0 [0 to 1]
Statistical Analysis 1: Comparison: Silicone (Coloplast Imajin Hydro) Ureteral Stent vs Non-silicone (Polyurethane/Percuflex) Ureteral Stent (Any Manufacturer); Test type: Superiority; p = 0.25, WinRatio, unmatched unstratified; WinRatio using unmatched method

8. Secondary Outcome: Abnormal Imaging Findings Within 60 Days
Description: Results reflect the participants whose imaging indicated either new or worsening hydronephrosis in the operative renal unit.
Time Frame: up to 60 days
Population: Only includes participants who received imaging (CT, US, and/or KUB) and were assessed for hydronephrosis within 60 days of URS
Measure: Count of Participants; unit: Participants
Arm/Group | Silicone (Coloplast Imajin Hydro) Ureteral Stent | Non-silicone (Polyurethane/Percuflex) Ureteral Stent (Any Manufacturer).
Number analyzed (Participants) | 37 | 47
Participants | 7 | 6
Statistical Analysis 1: Comparison: Silicone (Coloplast Imajin Hydro) Ureteral Stent vs Non-silicone (Polyurethane/Percuflex) Ureteral Stent (Any Manufacturer); Test type: Superiority; p = 0.44, Chi-squared

9. Secondary Outcome: Stone-free Rates Within 60 Days
Description: Results reflect the participants who had no residual renal stone following treatment based on postoperative imaging.
Time Frame: up to 60 days
Population: Only includes participants who received imaging (CT, US, and/or KUB) within 60 days of URS
Measure: Count of Participants; unit: Participants
Arm/Group | Silicone (Coloplast Imajin Hydro) Ureteral Stent | Non-silicone (Polyurethane/Percuflex) Ureteral Stent (Any Manufacturer).
Number analyzed (Participants) | 56 | 56
Participants | 33 | 32
Statistical Analysis 1: Comparison: Silicone (Coloplast Imajin Hydro) Ureteral Stent vs Non-silicone (Polyurethane/Percuflex) Ureteral Stent (Any Manufacturer); Test type: Superiority; p = 0.85, Chi-squared

ADVERSE EVENTS:
Time Frame: Up to 60 days
Arm/Group | Silicone (Coloplast Imajin Hydro) Ureteral Stent | Non-silicone (Polyurethane/Percuflex) Ureteral Stent (Any Manufacturer).
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/108
Serious Adverse Events (participants affected / at risk) | 3/107 | 2/108
Other Adverse Events (participants affected / at risk) | 11/107 | 10/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Silicone (Coloplast Imajin Hydro) Ureteral Stent (N=107) | Non-silicone (Polyurethane/Percuflex) Ureteral Stent (Any Manufacturer). (N=108)
Pyelonephritis (Renal and urinary disorders) | 0 | 1
Urinary Tract Infection (UTI) (Injury, poisoning and procedural complications) | 1 | 1
Hematuria (Renal and urinary disorders) | 1 | 1
Cystitis (Renal and urinary disorders) | 0 | 1
Flank Pain (Renal and urinary disorders) | 2 | 0
Nausea (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Silicone (Coloplast Imajin Hydro) Ureteral Stent (N=107) | Non-silicone (Polyurethane/Percuflex) Ureteral Stent (Any Manufacturer). (N=108)
Vulvovaginitis (Reproductive system and breast disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Infected and obstructing ureteral stone with AKI (Renal and urinary disorders) | 1 | 1
Stent Displacement (Renal and urinary disorders) | 3 | 0
Urinary Frequency (Renal and urinary disorders) | 2 | 1
Flank Pain (Renal and urinary disorders) | 5 | 5
Hematuria (Renal and urinary disorders) | 1 | 1
Fever (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 3 — Renal and Urinary Disorders
Nausea (Gastrointestinal disorders) | 2 | 2
Abdominal Pain (Gastrointestinal disorders) | 1 | 3
Fall resulting in arthroplasty (Musculoskeletal and connective tissue disorders) | 1 | 0
COVID (General disorders) | 1 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
PE without acure cor pulmonale (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructing Stone Fragment on Opposite Side (Renal and urinary disorders) | 1 | 0
Diarrhea and dehydration (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-12): https://cdn.clinicaltrials.gov/large-docs/10/NCT05026710/Prot_SAP_002.pdf